CLINICAL TRIAL: NCT00743873
Title: PRP Treatment for Medial Retinaculum Tear - Randomized-Double-Blind-Placebo Control Trail
Brief Title: Platelet-rich Plasma (PRP) Treatment for Medial Retinaculum Tear Post Medial Patellar Dislocation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Omer Mei-Dan, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4000
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Patella-Dislocation
Keywords: medial retinaculum tear s/p patella dislocation
MeSH Terms: conditions — Patellar Dislocation | interventions — Intercellular Signaling Peptides and Proteins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): saline
  Interventions: Drug: placebo
- 1 (Experimental): Plasma Rich in Growth Factors (PRGF)
  Interventions: Biological: Plasma Rich in Growth Factors (PRGF)

INTERVENTIONS:
Biological: Plasma Rich in Growth Factors (PRGF) — US guided IM injection 3-6mg
  Other Names: platelet-derived preparation rich in growth factors
  Arms: 1
Drug: placebo — injection of 6 cc of saline into injured area
  Other Names: saline 0.9% NaCl
  Arms: 2

SUMMARY:
To check the influence of injected platelet-rich plasma (PRP) on the healing of medial retinaculum and the redaction in recurrent dislocation of the patella.

DETAILED DESCRIPTION:
Autologous platelet-rich matrices may aid in the healing of ligaments & tendons by promoting and accelerating tissue healing because of the release of growth factors including transforming growth factor (TGF)-beta1 and platelet-derived growth factor (PDGF) from platelet alpha-granules.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years old
* first time patella dislocation

Exclusion Criteria:

* pregnancy
* mental or physical disabilities

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
redaction in healing time and recurrence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei Dan, Dr, Principal Investigator — Meir Medical Center
Locations (1):
- Meir medical center, Kfar Saba, Israel